CLINICAL TRIAL: NCT06973577
Title: A Phase 3b, Randomized, Double-blind, 8-week, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Centanafadine Once Daily Extended-release Capsules for the Treatment of Adults With Attention-deficit/Hyperactivity Disorder and Comorbid Anxiety
Brief Title: P3b Short-term Study of CTN in Patients With ADHD and Comorbid Anxiety
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 405-201-00180
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: ADHD; Anxiety; Generalized Anxiety; Social Anxiety Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Centanafadine QD XR fixed dose 328.8mg (Experimental)
  Interventions: Drug: Centanafadine

INTERVENTIONS:
Drug: Centanafadine — Centanafadine QD XR fixed dose 328.8mg
  Arms: Centanafadine QD XR fixed dose 328.8mg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Primary: To evaluate the efficacy of CTN in adults ages with ADHD and comorbid anxiety (AISRS) Key Secondary: To assess the efficacy of CTN in adults ages with ADHD and comorbid anxiety

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 18 and 65 years of age, inclusive.
2. Diagnosis of ADHD per the DSM-5-TR criteria and confirmed using the ACDS Version 1.2 at screening.
3. AISRS total score of ≥ 28 at baseline.
4. Diagnosis of GAD and/or SAD per DSM-5-TR criteria and confirmed using the MINI at screening.
5. HAM-A total score ≥ 20 at baseline.
6. CGI-S-ADHD and CGI-S-anxiety rating ≥ 4 at baseline.
7. Body mass index from 18.0 to 40.0 kg/m2 (inclusive).
8. Ability to provide written, informed consent prior to initiation of any trial-related procedures, and ability, in the opinion of the principal investigator, to comply with all the requirements of the trial.

Exclusion Criteria:

1. In the clinical opinion of the investigator, participant has not derived therapeutic benefit from 2 or more ADHD therapies of 2 different classes (eg, amphetamine and methylphenidate, or amphetamine and atomoxetine) given with an acceptable dose and duration during adulthood (aged 18 years or older).
2. In the clinical opinion of the investigator, participant has not derived therapeutic benefit from 2 or more anxiety therapies of 2 different classes (eg, selegiline and duloxetine, or buspirone and lorazepam) given with an acceptable dose and duration during adulthood (aged 18 years or older).
3. Current use of prohibited psychotropic medications that cannot be discontinued 2 weeks prior to randomization. Fluoxetine is prohibited within 28 days of randomization.
4. Participants who have started individual or group psychotherapy within the past 3 months prior to screening (ongoing psychotherapy that is not expected to change in frequency or type during the trial is permissible).
5. Any disorder that is the primary focus of treatment other than ADHD.
6. Participants with lifetime DSM-5-TR diagnosis of neurocognitive disorder, schizophrenia or any psychotic disorder, bipolar disorder, autism spectrum disorder, or personality disorders. Participants with current diagnosis of post-traumatic stress disorder, obsessive compulsive disorder, any substance use disorder, eating disorders, major depressive disorder; or other anxiety disorders such as panic disorder, agoraphobia, separation anxiety disorder, selective mutism, substance or medication induced anxiety, or due to medical condition, or specific phobia will be excluded.
7. Participant is, in the investigator's judgment, at significant risk for suicide. A participant with a Columbia-Suicide Severity Rating Scale (C-SSRS) ideation score of 4 or 5 within the last 6 months or participants who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) within the past year must be excluded.
8. Participants with a positive UDS for illicit drugs at screening or baseline. Participants with a positive drug test at screening for ADHD or anxiety medications including methylphenidate, or amphetamines, may continue while undergoing the required washout. Participants with a positive drug test at baseline for ADHD or anxiety medications are excluded. A positive drug test at baseline for drugs of abuse, including cannabis, unless all of the following cannabis specific conditions are met:

   1. No DSM-5-TR diagnosis of cannabis use disorder within the past 12 months;
   2. If per investigator's judgement, cannabis use will not compromise safety, efficacy assessments or protocol compliance.
   3. Participant agrees to maintain their consistent use pattern throughout the trial
   4. Participant agrees to refrain from cannabis use within 12 hours of trial visits.
9. Participants with evidence of current substance use disorder or history in the past 12 months.
10. Participants with epilepsy, a history of epilepsy, or a history of seizure, except for a single childhood febrile seizure, a single seizure post brain injury, or a single seizure due to alcohol withdrawal.
11. Participants who are partially hospitalized or receiving inpatient care or have any other medical or physical condition(s) that, in the opinion of the investigator, may prevent the participant from completing the trial or would go against the participant's best interest with participation in the trial. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. This would also include most bariatric surgeries, with the only exception being those where there has been no breach of the gastrointestinal wall (ie, uncomplicated lap band surgery) AND no sign of malabsorption.
12. The following laboratory test and ECG results are exclusionary at screening:

    1. Platelets ≤ 75,000/mm3
    2. Hemoglobin ≤ 9 g/dL
    3. Neutrophils, absolute ≤ 1000/mm3
    4. AST > 2 × upper limit of normal
    5. ALT > 2 × upper limit of normal
    6. Creatinine ≥ 2 mg/dL
    7. HbA1c ≥ 7%
    8. QTcF ≥ 450 msec for males or ≥ 470 msec for females
    9. Abnormal free thyroxin (T4), unless discussed with and approved by the medical monitor (Note: free T4 is measured only if result for thyroid stimulating hormone [TSH] is abnormal)
13. Participants presenting with, or having a history of, uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg) or symptomatic hypotension, or orthostatic hypotension which is defined as a decrease of ≥ 30 mmHg in systolic blood pressure or a decrease of ≥ 20 mmHg in diastolic blood pressure after at least 3 minutes standing compared with the previous supine blood pressure, or development of symptoms.
14. Participants with a history of any prior exposure to centanafadine.
15. Participants who have participated in other clinical trials involving investigational drugs within 180 days prior to screening or who have participated in more than 2 interventional clinical trials involving investigational drugs within the past year.
16. Participants of childbearing potential who are breast-feeding and/or have a positive pregnancy test result prior to receiving IMP.
17. Participants of reproductive potential / POCBP who do not agree to practice 2 different effective and/or highly effective methods of birth control or remain fully abstinent from sexual activity with the potential for conception, per the guidelines in Section 10.3.
18. Participants who do not agree to refrain from donating sperm or eggs from trial screening through 90 days for sperm and 30 days for eggs after the last dose of IMP.
19. Participants who have an allergy to the IMP or any component of the IMP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-10-04 (Estimated)

PRIMARY OUTCOMES:
Change in Adult Investigator Symptom Rating Scale (AISRS) | Baseline to Week 8
  The AISRS is an 18-item clinician rating scale to evaluate individual ADHD symptoms on a scale of 0 (none) to 3 (severe). The total sum ranges from 0 (no ADHD symptoms) to 54 (extremely severe ADHD symptoms). Negative change from Baseline indicates improvement.

SECONDARY OUTCOMES:
Change in Hamilton Anxiety Rating Scale (HAM-A) | Baseline to Week 8
  The HAM-A consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a 5-point scale, ranging from 0 = not present to 4 = very severe. Negative change from Baseline indicates improvement.

CONTACTS AND LOCATIONS:
Locations (47):
- United States (46):
  - Clinical Research Site #017 - Harmonex Neuroscience Research, Dothan, Alabama
  - Clinical Research Center #033 - Woodland International Research Group, Little Rock, Arkansas
  - Clinical Research Center #048 - Woodland Research Northwest, Rogers, Arkansas
  - Clinical Research Site #052 - Leading Edge Research LA, LLC, Encino, California
  - Clinical Research Center #008 - Long Beach Clinical Trial Services Inc., Long Beach, California
  - Clinical Research Site #008 - Long Beach Clinical Trial Services Inc., Long Beach, California
  - Clinical Research Site #011 - NRC Research Institute, Orange, California
  - Clinical Research Center #042 - Anderson Clinical Research, Redlands, California
  - Clinical Research Site #037 - Cenexel CIT IE (Clinical Innovations Inc), Riverside, California
  - Clinical Research Site #039 - California Neuroscience Research, LLC, Sherman Oaks, California
  - Clinical Research Site #038 - Sunwise Clinical Research, Walnut Creek, California
  - Clinical Research Site #030 - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Clinical Research Site #045 - Research Center for Clinical Studies, Norwalk, Connecticut
  - Clinical Research Center #035 - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Research Site #005 - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Research Site #046 - ARSN-Largo CRU, Largo, Florida
  - Clinical Research Site #010 - Meridien Research/Accel Clinical, Maitland, Florida
  - Clinical Research Site #015 - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Research Site #006 - CNS Healthcare Orlando, Orlando, Florida
  - Clinical Research Site #019 - Segal Trials Innovatice Clinical Research, Inc., Tamarac, Florida
  - Clinical Research Site #004 - CenExel iResearch, LLC, Decatur, Georgia
  - Clinical Research Site #002 - Psych Atlanta, PC, Marietta, Georgia
  - Clinical Research Center #032 - CenExel iResearch, LLC, Savannah, Georgia
  - Clinical Research Center #056 - Research Works INC., New Orleans, Louisiana
  - Clinical Research Site # 027 - Copley Clinical, Boston, Massachusetts
  - Clinical Research Center #022 - Boston Clinical Trials - Alcanza Clinical Research, LLC, Boston, Massachusetts
  - Clinical Research Site #025 - Adams Clinical, Watertown, Massachusetts
  - Clinical Research Site #016 - Clinical Research of Southern Nevada, LLC, Las Vegas, Nevada
  - Clinical Research Center #031 - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Clinical Research Site #026 - Neurobehavioral Research Inc, Cedarhurst, New York
  - Clinical Research Site #021 - The Medical Research Network, LLC, New York, New York
  - Clinical Research Site #028 - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - Clinical Research Site #047 - Insight Clinical Trials, Independence, Ohio
  - Clinical Research Site #009 - Paradigm Research Professionals LLC, Oklahoma City, Oklahoma
  - Clinical Research Site #023 - Summit Headlands LLC, Portland, Oregon
  - Clinical Research Site # 029 - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Clinical Research Site #014 - Suburban Research Associates, Media, Pennsylvania
  - Clinical Research Center #059 - Adams Clinical Philadelphia, Philadelphia, Pennsylvania
  - Clinical Research Center #034 - Coastal Carolina Research Center, North Charleston, South Carolina
  - Clinical Research Site #001 - CNS Healthcare - Memphis, Memphis, Tennessee
  - Clinical Research Site #013 - Donald J. Garcia, Jr. MD., PA, Austin, Texas
  - Clinical Research Site #020 - Houston Clinical Trials LLC, Bellaire, Texas
  - Clinical Research Site #003 - FutureSearch Trials of Dallas LP, Dallas, Texas
  - Clinical Research Site #012 - Clinical Trials of Texas, San Antonio, Texas
  - Clinical Research Site #036 - Grayline Research Center, Wichita Falls, Texas
  - Clinical Research Site #024 - Core Clinical Research, Everett, Washington
- Clinical Research Center #062 - Research Works - San Juan, Guaynabo, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the result of this study will be shared with researchers to achieve aims pre-specified in a methodology sound research proposal.
  Supporting Information:
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: http://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com